CLINICAL TRIAL: NCT05307770
Title: Randomized, Double-Blind, Cross-Over Study Comparing the Efficacy of Immediate and Extended-Release Melatonin as a Supplement Affecting the Sleep Cycle in Patients With Parkinson Disease and Rapid Eye Movement Sleep Behavior Disorder
Brief Title: Extended-Release Melatonin in Patients With Rapid Eye Movement Sleep Behavior Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emir Festic, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-003326
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Rapid Eye Movement Sleep Behavior Disorder; Parkinson Disease
MeSH Terms: conditions — REM Sleep Behavior Disorder; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Release Melatonin, Then Extended Release Melatonin (Experimental): Subjects will receive immediate release melatonin 5 mg orally at 9 pm every night for 4 weeks. After a washout period of 2 weeks, they then receive extended release melatonin 5 mg orally at 9 pm every night for 4 weeks.
  Interventions: Dietary Supplement: Immediate Release Melatonin; Dietary Supplement: Extended Release Melatonin
- Extended Release Melatonin, Then Immediate Release Melatonin (Experimental): Subjects will receive extended release melatonin 5 mg orally at 9 pm every night for 4 weeks. After a washout period of 2 weeks, they then receive immediate release melatonin 5 mg orally at 9 pm every night for 4 weeks.
  Interventions: Dietary Supplement: Immediate Release Melatonin; Dietary Supplement: Extended Release Melatonin

INTERVENTIONS:
Dietary Supplement: Immediate Release Melatonin — 5 mg orally every night at 9 pm for 4 weeks
Dietary Supplement: Extended Release Melatonin — 5 mg orally every night at 9 pm for 4 weeks

SUMMARY:
The purpose of this research is to compare the efficacy of immediate versus extended-release melatonin as a supplement affecting the sleep cycle in patients with Parkinson disease and Rapid Eye Movement Sleep Behavior Disorder.

DETAILED DESCRIPTION:
Enrolled patients with Parkinson disease and previously diagnosed rapid eye movement sleep behavior disorder, who are being treated at Mayo Clinic in Florida, will be randomized to receive either immediate-release melatonin or extended-release melatonin and then will be crossed over to receive the opposite intervention. The study will consist of two treatment periods of 4 weeks separated by a washout period of 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease and rapid eye movement sleep behavior disorder.
* Patient registered to Parkinson's disease database of Mayo Clinic Florida.

Exclusion Criteria:

* Patients who are using other sleep aids or medications (Clonazepam).
* Patients who are not willing to undertake 1 week of washout period.
* Patients who do not sign a consent for research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Change in sleep cycle | Baseline and 4 weeks
  Assessed by the self-reported modified Mayo Sleep questionnaire (MSQ) which consists of 8 questions related to sleep behavior in the past month.

CONTACTS AND LOCATIONS:
Overall Officials: Emir Festic, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States